CLINICAL TRIAL: NCT07300553
Title: Impact Of The Gut Microbiota On Host Cells Energy Metabolism in Health And In Inflammatory Bowel Disease
Acronym: ENERGISED
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: INSERMUMR938 (Unknown); CRB SAT APHP.SU Saint-Antoine hospital (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: APHP221107
Record Dates: First submitted 2025-12-10; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: IBD; Crohn Disease; Ulcerative Colitis (UC)
Keywords: Energy Metabolism; Gut Microbiota; Healthy volunteers; Patients with IBD; SCENITH analysis; Antimicrobial treatment; Inulin; Biological collection
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative | interventions — Vancomycin; Amphotericin B; Inulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy volunteers (Experimental): Healthy volunteer will be seen by a physician from the CRC-Est in LRIPH Saint-Antoine to verify their eligibility and collect their written consent. The baseline visit (V1) takes place within 4 weeks after the inclusion visit (V0). Antimicrobial treatment will be provided to the participant (7/8 days treatment). V2 takes place 7 days after baseline visit after the antimicrobial treatment For each visit (V1 and V2) the participants will be seen by a research physician and nurse after an overnight fast. Blood sample (for SCENITH analysis) will be perfomed. Then, participants will receive a standard breakfast with 10g 13C-labeled inulin, which serves as a model fermentable substrate. Blood samples (8mL) will be then collected every hour between 2 and 10h after consumption of the breakfast. All urines and stool samples emitted during the day D0 will be collected (and time recorded). Follow up at D2 to D3 post V1 will be done by a phone interview by CRT or nurse with the help and validati
  Interventions: Drug: Vancomycin /Amphotericin B (Fungizone®) /Gentamicine 80 mg
- Patients with IBD (Experimental): IBD patients will be seen by a gastroenterologist from the Gastroenterology department of the Saint-Antoine hospital or physician from the CRC-Est in LRIPH or the gastroenterology department of Saint Antoine to verify their eligibility, and collect their written consent during a usual follow up visit. The baseline visit (V1) takes place within 4 weeks after the inclusion visit (V0). The patients will be seen by a research physician and nurse after an overnight fast. Blood sample (for SCENITH analysis) will be perfomed. Then, participants will receive a standard breakfast with 10g 13C-labeled inulin, which serves as a model fermentable substrate. Blood samples (7mL) will be then collected every hour between 2 and 10h after consumption of the breakfast. All urines and stool samples emitted during the day D0 will be collected (and time recorded). The patient will also receive a kit for fecal collection at home to be done the day before v1.
  Interventions: Dietary Supplement: Inulin/Inulin C13

INTERVENTIONS:
Drug: Vancomycin /Amphotericin B (Fungizone®) /Gentamicine 80 mg — 7 days treatment taken over 8 calendar days).
  The first intake will take place just before leaving the hospital on the evening of day 0. A precise schedule will be provided for the antibiotics intakes, with the last intake in the afternoon on day 7 (on day 7, only 3 intakes of antibiotics: morning, noon and afternoon):
  Vancomycin VIATRIS 500 mg for injection or oral administration Dose: 250mg x4 daily orally Amphotericin B (Fungizone®) Bottle 10% (4000mg/40ml) oral solution Dose 500mg x4 (20ml) daily orally Gentamycine 80 mg/2 ml solution (hospital compounding) Dose 80mg x4 daily orally
  Arms: Healthy volunteers
Dietary Supplement: Inulin/Inulin C13 — - INULIN ; food grade inulin from Chicory (2% labelled with 13C) at H0 on day 0 (v1) and day 7 (v2) for healthy adults and day 0 (v1) only for patients with IBD.
  Arms: Patients with IBD

SUMMARY:
Inflammatory Bowel Disease (IBD) often leads to poor disease control and reduced quality of life. Changes in the gut microbiota may disrupt the energy metabolism of immune cells, contributing to IBD.

This study will examine how gut microbiota affects immune cell metabolism in healthy adults and IBD patients. Healthy volunteers will be tested before and after a short antibiotic treatment, while IBD patients will be tested once.

Energy metabolism will be measured using SCENITH, a method that analyzes metabolic activity in blood immune cells.

Participants will also receive a special form of fiber (13C-labeled inulin) to track how gut bacteria break down and use this nutrient. Blood, urine, and stool samples will be analyzed to follow the metabolic fate of inulin. DNA and RNA from stool will be studied to identify which bacteria metabolize the labeled fiber.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteer

1. Age ≥ 18 years and < 50 years
2. 17 kg/m² < body mass index < 25 kg/m² (microbiota modified based on BMI, (Le Chatelier et al., 2013)
3. For women, female of child-bearing age with an active contraception (hormonal, intrauterine device, bilateral tubal occlusion, sexual abstinence*) and this during at least the period of treatment (up to v2) *Sexual abstinence is defined as refraining from heterosexual intercourse from providing consent until V3. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the participant

   * A woman is considered of childbearing potential, i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH), level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient
4. Regular bowel movement defined as at least 1 stool every other day and maximum 3 stools per day
5. Patient with health insurance (AME except)
6. Informed Written consent Patient with IBD

<!-- -->

1. Age ≥ 18 years and < 50 years
2. Crohn's Disease (Excepting disease involving only the upper GI tract) or ulcerative colitis (excepting disease involving only the rectum), according to the Lennard-Jones criteria for at least 6 months (15 patients with Crohn's disease and 15 with ulcerative colitis will be recruited)
3. Patient in steroid-free clinical remission for at least 6 months (for Crohn's disease: CDAI <150 the week before inclusion, for ulcerative colitis: Partial Mayo Clinic score of 0 or 1).
4. 17 kg/m² < body mass index < 25 kg/m²
5. Female of child-bearing age with an active contraception. Efficient contraception include oral contraception, intrauterine devices hormonal device, intrauterine hormone-releasing system, sterilization method and other forms of contraception with failure rate <1%)

   ** A woman is considered of childbearing potential, i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy.

   A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient
6. Regular bowel movement defined as at least 1 stool every other day and maximum 3 stools per day
7. Patient with health insurance (AME except)
8. Informed Written consent

Non inclusion Criteria:

Healthy volunteers

1. Significant chronic disease and particularly chronic gastrointestinal diseases, type 1 and type 2 diabetes, renal alteration
2. Curative long-term treatment
3. Pregnant or breastfeeding women** ** A woman is considered of childbearing potential, i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy.

   A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.
4. blood donation in the 3 months before the study
5. Taking antibiotic or antifungal (oral) in the previous 3 months before planned day 0 (V1)
6. probiotics in the month preceding day 0 (V1),
7. consumption of a low-calorie diet or any other special diet (except vegetarian) in the month before day 0
8. abdominal surgery in the past (except for appendectomy)
9. allergy against the antibiotics and antifungal treatment used in this study or to their excipients
10. contra-indications to the administration of gentamicin (refer to SmPC)
11. Participation in any other interventional study
12. Patients under legal protection Patients with IBD

<!-- -->

1. Pregnant or breastfeeding women
2. blood donation in the 3 months before the study
3. Taking antibiotic or antifungal (oral) in the previous 3 months before planned day 0
4. probiotics in the month preceding day 0 and during the study,
5. Ileal resection > 50cm or colectomy
6. Diagnosis of Crohn's disease restricted to the upper gastrointestinal tract (oesophagus, stomac, duodenum, jejunum)
7. Diagnosis of ulcerative colitis restricted to the rectum.
8. Current stoma (Ileostomy or a colostomy) or stoma in the last 6 months or any other intra-abdominal surgery within 3 months prior to inclusion
9. Participation in any other interventional study
10. Patients under legal protection

Exclusion Criteria:

Healthy volunteers :

* Clinically significant abnormal serum/ plasma levels of electrolytes, creatinine, liver enzymes, thyroid stimulating hormone or blood cell count at the biological check-up of the visit v0 (screening and inclusion)
* Infectious episode requiring antimicrobial treatment since V0
* Severe diarrhea (increase of seven or more stools per day over baseline)

Patients with IBD - Infectious episode requiring antimicrobial treatment since V0

- IBD flare

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Evaluate the impact of the gut microbiota, and of its alteration in inflammatory bowel disease, on peripheral immune cells energy metabolism | Healthy volunteers : 7 days/ IBD patients : 1 day
  Energy metabolism of major immune cell types for peripheral blood will be assessed on a blood sample
  * For healthy adults, this analysis will be performed on blood sample at day 0 (v1, before antimicrobial treatment onset) and at day 7 (v2, last day of the antimicrobial treatment).
  * For patients with IBD this analysis will be performed on blood sample at day 0 (v1).
  The energy metabolism will be assessed by single-cell energetic metabolism by profiling translation inhibition (SCENITH) approach (Argüello et al., 2020). SCENITH is a flow cytometry-based approach allowing to functionally profile energy metabolism with single-cell resolution from a simple blood sample

SECONDARY OUTCOMES:
Evaluate the impact of the gut microbiota and its alteration in inflammatory bowel disease on the fate of microbiota-derived carbon sources in host cells | Healthy volunteers : 7 days/ IBD patient : 1 day
  we will use a strategy based on stable isotope probing (SIP). The participants will receive orally food grade inulin from Chicory (2% labelled with 13C) at H0 on day 0 (v1) and day 7 (v2) for healthy adults and day 0 (v1) only for patients with IBD. The incorporation of 13C in metabolites will then be assessed Targeted (TCA cycle and glycolysis intermediates and fatty acids) and untargeted metabolomics will be performed on blood samples obtained every hour from 2 h to 10 h post inulin intake on day 0 (v1) and day 7 (v2) for healthy adults and day 0 (v1) only for patients with IBD.
  * Similar analysis will be performed on each urine samples emitted during day 0 (v1) and day 7 (v2) for healthy adults and day 0 (v1) for patients with IBD.
  * Similar analysis will be performed on each fecal samples emitted during day 0 (v1) and day 7 (v2) for healthy adults and day 0 (v1) for patients with IBD. Stool emitted on day 1 and on day 8 will be also collected for analysis.
Identify the intestinal bacteria involved in this process | Healthy volunteers : 7 months and 8 days/IBD patient : 4 weeks and 2 days
  we will use SIP-DNA and SIP-RNA sequencing approaches (Fortunato and Huber, 2016; Neufeld et al., 2007; Ziels et al., 2018). DNA and RNA will be extracted from each fecal samples obtained (see above). Labeled DNA/RNA will be separated by density gradient centrifugation. The "heavier" labeled nucleic acid fractions, corresponding to microorganisms that metabolized labeled inulin and incorporated labeled atoms into their nucleic acids, will undergo 16s and/or shotgun sequencing to identify the inulin-metabolizing taxa.

CONTACTS AND LOCATIONS:
Overall Officials: Harry SOKOL, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Gastroenterology Department Saint Antoine Hospital,, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided